CLINICAL TRIAL: NCT06849297
Title: Effectiveness of Aromatherapy in Reducing Anxiety and Pain Perception in Women During Childbirth
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Andrzej Frycz Modrzewski Krakow University (Other)
Responsible Party: Principal Investigator, Renata Bakalarz, doctor, Andrzej Frycz Modrzewski Krakow University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: KBKA/18/O/2024
Record Dates: First submitted 2025-02-24; First posted 2025-02-27 (Actual); Last update posted 2025-02-27 (Actual); Status verified 2025-02

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Aromatherapy Group (Intervention Arm) (Experimental): Participants will receive aromatherapy during labor, using essential oils as recommended by medical staff and based on individual preferences. The laboring woman will choose the type of oil and method of application. Before use, a midwife will inform her about the properties and application methods of essential oils.
  Possible aromatherapy applications during labor:
  * Diffusion: Dispersing essential oils in the air using a diffuser to create a relaxing atmosphere. Oils like lavender, geranium, and mandarin may help reduce tension and anxiety.
  * Massage: Essential oils mixed with a carrier oil (e.g., coconut or almond) can be used for gentle massage of the back, arms, or feet to ease muscle tension and discomfort.
  * Infused cloths: Essential oil-soaked cloths or compresses can be used for inhalation. The woman can hold the cloth near her nose during contractions to aid relaxation.
  The medical staff will offer different essential oils depending on the woman's preferences.
  Interventions: Behavioral: Aromatherapy during labor
- Control Group (Standard Care Arm) (No Intervention): Participants in this group will receive standard obstetric care without the use of aromatherapy.
  All routine childbirth procedures will be applied according to hospital protocols.
  This arm serves as the baseline for comparing the effectiveness of aromatherapy against standard care in terms of pain management, anxiety reduction, and childbirth satisfaction.
  Randomization will ensure equal distribution of participants into both arms to enable an objective comparison of the outcomes associated with aromatherapy versus standard obstetric care.

INTERVENTIONS:
Behavioral: Aromatherapy during labor — Use of essential oils (diffusion, massage, or infused cloths) during labor to promote relaxation and pain relief.
  Arms: Aromatherapy Group (Intervention Arm)

SUMMARY:
Study Summary

Objective of the StudyThis study aims to evaluate the effects of aromatherapy on women's childbirth experiences, particularly in reducing anxiety, alleviating pain, and increasing overall satisfaction with labor. The research seeks to explore whether aromatherapy can serve as an effective, non-pharmacological method to improve comfort during childbirth.

Research QuestionDoes the use of aromatherapy during labor reduce pain intensity, lower anxiety levels, and enhance maternal satisfaction compared to standard obstetric care?

HypothesisIt is hypothesized that the use of aromatherapy during labor helps to decrease anxiety, lessen labor pain, and improve the overall birth experience without negatively affecting the health of the mother or newborn.

Brief Description of the StudyThis study is a randomized controlled clinical trial conducted at the Stefan Żeromski Specialist Hospital in Kraków. It will include women who are delivering vaginally between 37-42 weeks of gestation. Participants will be randomly assigned to either a group receiving aromatherapy (using essential oils such as lavender, clary sage, and lemon) or a control group receiving standard obstetric care without aromatherapy.

The effectiveness of aromatherapy will be assessed based on pain perception, anxiety levels, labor duration, and newborn condition. The study aims to provide scientific evidence on the benefits of aromatherapy in labor, potentially contributing to its broader adoption in maternity care.

DETAILED DESCRIPTION:
Study Summary Study Objective The objective of this study is to evaluate the impact of aromatherapy on women's childbirth experiences, including anxiety reduction, pain perception, and overall satisfaction with the delivery process. Given the increasing interest in non-pharmacological pain and stress relief methods during labor, this study aims to provide reliable scientific data on the effectiveness of aromatherapy as a supportive method for laboring women.

Research Question Does the use of aromatherapy during labor reduce labor pain, lower anxiety levels, and improve overall satisfaction with the childbirth experience compared to standard obstetric care? Research Hypothesis It is hypothesized that the use of aromatherapy during labor leads to reduced anxiety levels, decreased intensity of labor pain, and increased satisfaction with the childbirth experience, without adverse effects on maternal and neonatal health.

Study Description

This is a randomized controlled clinical trial conducted at the Labor and Delivery Ward of the Stefan Żeromski Specialist Hospital in Kraków. Women delivering vaginally between 37-42 weeks of gestation will be included. Participants will be randomly assigned to one of two groups:

* Experimental Group - use of aromatherapy during labor, including diffusion of essential oils, inhalation, or massage with patient-selected oils (e.g., lavender, clary sage, lemon, geranium, peppermint).
* Control Group - standard obstetric care without the use of aromatherapy. Methods for Evaluating Aromatherapy Effectiveness
* Pain assessment using the Visual Analogue Scale (VAS).
* Anxiety level assessment using the Childbirth Anxiety Questionnaire (KLP II).
* Analysis of childbirth satisfaction using the Childbirth Experience Questionnaire (QACE).
* Evaluation of the impact of aromatherapy on labor duration and perineal incision rates.
* Neonatal assessment using the Apgar score and determining the need for hospitalization in the Neonatal Pathology Unit.
* Postpartum depression assessment two weeks after birth using the Edinburgh Postnatal Depression Scale (EPDS).

Detailed Study Description Study Design The study is designed as a randomized controlled clinical trial (RCT) with double-blinded allocation to study groups. Randomization will be performed using a computer algorithm, and group assignment will remain concealed until the intervention begins.

Study Procedure The study is divided into three phases: the preliminary phase, the main study phase, and the data analysis phase.

* Preliminary Phase - Adaptation of research tools to Polish conditions, pilot tests, and training of medical personnel.
* Main Study Phase - Conducting the study according to protocol, participant enrollment, and data collection.
* Analysis Phase - Statistical data analysis and interpretation of results. Intervention In the experimental group, doTERRA essential oils will be used, selected based on patient preferences and medical indications. Possible application methods include diffusion, inhalation, and massage.

Data Collection Methods

Data will be collected at multiple stages:

* Upon study enrollment (demographic questionnaire, medical history).
* During labor (VAS pain assessment, KLP II anxiety measurements).
* After childbirth (QACE childbirth satisfaction assessment, neonatal Apgar scores).
* Two weeks postpartum (EPDS postpartum depression assessment). Study Significance The results are expected to provide scientific evidence on the effectiveness of aromatherapy in reducing labor pain and anxiety. The study findings may contribute to the widespread implementation of aromatherapy as a standard supportive method in obstetric care.

ELIGIBILITY:
Inclusion Criteria:

* Female participants.
* Minimum age of 18 years.
* Pregnant women between 37 and 42 weeks of gestation.
* Planning a vaginal delivery.
* In overall good health, without pregnancy-related complications.
* Willing to provide informed consent for participation in the study.
* No history of high-risk pregnancy.
* Ability to understand the study procedures and follow instructions.

Exclusion Criteria:

* Severe maternal health conditions that may affect labor outcomes.
* High-risk pregnancy requiring medical interventions.
* Presence of fetal congenital anomalies.
* Decision to receive epidural or other pharmacological pain relief.
* Need for medical intervention during labor (e.g., cesarean section, forceps, vacuum extraction).
* Known allergies or adverse reactions to essential oils.
* Inability to provide informed consent due to cognitive impairment or language barriers.
* Presence of chronic respiratory conditions that may be affected by inhaled essential oils.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Only female participants are eligible for this study, as it focuses on the effects of aromatherapy during labor and childbirth, which are exclusive to women.
Enrollment: 300 (Estimated)
Dates: Start 2025-02-17 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Pain intensity during labor measured by Visual Analog Scale (VAS) | At cervical dilation of 3 cm, 6 cm, and 9 cm,
  Pain intensity will be assessed using the Visual Analog Scale (VAS), where 0 represents no pain and 10 represents the worst pain imaginable. Measurements will be taken multiple times: at 3 cm, 6 cm, and 9 cm cervical dilation, Pain scores will be compared between the aromatherapy and control groups.

SECONDARY OUTCOMES:
MMaternal anxiety during labor measured by Childbirth Anxiety Questionnaire (KLP II) | 1 hour after the start of aromatherapy (or at the same time point in the control group without aromatherapy).
  Anxiety levels during labor will be assessed using the Childbirth Anxiety Questionnaire (KLP II). Measurements will be taken approximately 1 hour after the start of aromatherapy in the intervention group. In the control group, anxiety levels will be assessed at the same time point without aromatherapy. Anxiety scores will be compared between both groups.
Maternal satisfaction with childbirth experience measured by QACE (Questionnaire for Assessing the Childbirth Experience) | 2 hours postpartum
  Overall satisfaction with the childbirth experience will be assessed using the QACE questionnaire. Measurements will be taken 2 hours after birth and compared between the aromatherapy and control groups.
Postpartum depression symptoms assessed using the Edinburgh Postnatal Depression Scale (EPDS) | 2 weeks postpartum
  The Edinburgh Postnatal Depression Scale (EPDS) will be used to assess postpartum depression symptoms. A higher score indicates a greater likelihood of postpartum depression. Data will be collected 2 weeks postpartum via an online questionnaire.

CONTACTS AND LOCATIONS:
Locations (1):
- Stefan Żeromski Specialist Hospital in Kraków, Krakow, Poland

IPD SHARING:
Plan to Share IPD: Undecided
Currently, we have not made a final decision about sharing individual participant data (IPD). The decision to share data will depend on factors such as obtaining ethical approvals, participant consent for data sharing, as well as ensuring adequate privacy protection and data anonymization procedures. The final determination will be made in accordance with institutional policies and ethical standards following the completion of the study.